CLINICAL TRIAL: NCT01078103
Title: Corneal Endothelial Changes Associated With Phacoemulsification in Diabetes
Brief Title: Corneal Endothelial Changes Associated With Phacoemulsification in Diabetes Mellitus Type II
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Allan Storr-Paulsen, Frederiksberg University Hospital
Other Study IDs: J.nr.2005-41-4933
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes; Cataract
Keywords: Diabetes Mellitus; cornea endothelium; cell loss; cataract surgery
MeSH Terms: conditions — Diabetes Mellitus; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Some studies indicated that the diabetic corneal endothelium is morphologically abnormal and may be at risk in any intraocular surgical procedure, while others showed no significant differences between diabetic and non-diabetic corneal endothelium.The purpose of this study is to investigate the differences in corneal endothelial cell density and morphology in diabetic patients and normal patients after phacoemulsification with intraocular lens implantation.To investigate if haemoglobin A1c can be used as a predictor of corneal endothelial cell changes after phacoemulsification.

DETAILED DESCRIPTION:
Some studies indicated that the diabetic corneal endothelium is morphologically abnormal and may be at risk in any intraocular surgical procedure, while others showed no significant differences between diabetic and non-diabetic corneal endothelium.The purpose of this study is to investigate the differences in corneal endothelial cell density and morphology in diabetic patients and normal patients after phacoemulsification with intraocular lens implantation.To investigate if haemoglobin A1c can be used as a predictor of corneal endothelial cell changes after phacoemulsification.

Specular microscopy photos will be taken pre-. and 3 month postoperatively. Cellular parameters will be compared between the two groups prior and post surgery. Clinical significant difference is defined as 1 SD (300 cell/mm2)

ELIGIBILITY:
Inclusion Criteria:

* Cataract, diabetes

Exclusion Criteria:

* Corneal disease
* Uveitis
* Previous intraocular surgery and diabetes type I

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 typoe II diabetic and 30 non diabetic undergoing catarct surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan V Storr-Paulsen, MD, Study Director — Frederiksberg University Hospital
Locations (1):
- Frederiksberg Hospital, Copenhagen, Denmark